CLINICAL TRIAL: NCT05865951
Title: Long-term Comparative Effects of Isometric and Isotonic Global Neck Muscles Strengthening Exercise Program on Pain, Range of Motion, Strength, Function, and Quality of Life in Patients With Chronic Mechanical Neck Pain.
Brief Title: Comparison of Isometric and Isotonic Strengthening Exercises in Chronic Neck Pain Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0117
Record Dates: First submitted 2023-04-18; First posted 2023-05-19 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chronic neck pain and isometric exercises group: (Experimental): Group A performed exercises for 12 weeks. Participants performed isometric exercises along with conventional physical therapy treatment ( thermotherapy, manual mobilisation of cervical spine and trigger point therapy). All exercises were performed for 3 sessions per week for a period of 12 weeks.
  Interventions: Other: Isometric Exercises
- chronic neck pain and isotonic group (Active Comparator): Group B performed exercises for 12 weeks. Participants performed isotonic exercises along with conventional physical therapy treatment ( thermotherapy, manual mobilisation of cervical spine and trigger point therapy). All exercises were performed for 3 sessions per week for a period of 12 weeks.
  Interventions: Other: Isotonic Exercises

INTERVENTIONS:
Other: Isometric Exercises — Isometric (same length) strengthening exercises of the neck muscles will be performed.
  Arms: chronic neck pain and isometric exercises group:
Other: Isotonic Exercises — Isotonic strengthening exercises for the neck muscles will be performed.
  Arms: chronic neck pain and isotonic group

SUMMARY:
Study will be a Randomized clinical trial to check the effects of isometric and isotonic strength training exercises on patients with chronic neck pain. The data will be collected in a hospital setting where patients of chronic mechanical neck pain will be screened out for the fulfillment of eligibility criteria of this study. After being eligible for this study their baseline outcome measures will be measured using Numeric pain rating scale, neck disability index, goniometer, dynamometer and short form 36 survey. Then they will be divided into two groups namely group A receiving isometric exercises with conventional treatment and group B receiving isotonic exercises with conventional treatment. Here conventional treatment includes thermotherapy, manual mobilisation of cervical and thoracic and trigger point therapy which will be a common treatment for both groups. The outcome measures will be measured later at 4th,8th and 12th week.

DETAILED DESCRIPTION:
Chronic neck pain is a burden to health globally and is the major reason behind years of disability. This is due to the higher prevalence, persistence and recurrence.It is a frequent reason for visit to physical therapist or a physician. It is the major health concern for society these days with highest recurrence rate combined with its chronicity. The overall worldwide prevalence for it is 16.7% to 75.1%. There is scarce knowledge of use of isotonic neck muscles strengthening in clinical trials. Moreover the literature has not satisfied the long term effects of isometric and isotonic strength training exercises of cervical muscles on improving the health related quality of life and restoring the normal function of cervical spine.

The findings of current study will help to establish long term effects of isometric and isotonic strengthening exercises on pain, strength, function and quality of life in chronic mechanical neck pain patients.

Neck strength training exercises have shown to reduce neck muscle injuries in sports.Neck strength training has also proved beneficial in reducing neck pain as part of training.

The static muscle contractions of neck muscles of patient being seated with the resistance of palm of physiotherapist being standing will be performed in six cervical movements i.e. flexion, extension, right lateralflexion, left lateral flexion, right rotation, left rotation.

The dynamic muscle contractions of neck muscles will be performed using thera-band for resistance tied on the wall for all six movements of cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* No discrimination against gender
* Age group 25-55 years
* Complain of chronic mechanical neck pain for more than 3 months

Exclusion Criteria:

* Spinal cord injury
* Malignancy
* Cervical fracture
* Any bony or soft tissue systemic disease
* Ankylosis spondylitis
* Craniovertebral disorders
* Any cervical deformity

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS): | up to 12 weeks
  It is a unidimensional outcome measure that is used for measuring intensity of chronic pain. It is a verbally administered scale rating from 0 to 10 where 10 quantifies worse pain intensity and 5 as a moderate intensity. The simplicity in pain scoring makes it a reliable scale with reliability 0.96 in literate and 0.95 in illiterate patients whereas validity ranges from 0.86 to 0.95.
Universal GONIOMETER for Range of Motion | up to 12 weeks
  It is the device used for measuring range of motion of joints. One of the type of goniometer to be used in this study is universal goniometer with two arms, one arm is maintained at neutral position whereby the other arm moves with the moving part of body. The inter-observer reliability remains at 0.99 whereas validity being 0.97
Hand-Held DYNAMOMETER for muscle strength measurement | up to 12 weeks
  Dynamometer is a hand-held device used to measure thestrength of muscles. It is to be placed as a resistance in the movement to quantify the muscle strength into force unit. It has reliability from 0.94 to 0.97.
NECK DISABILITY INDEX (NDI): | up to 12 weeks
  It is a function specific questionnaire designed to measure thelevel of disability and restriction in activities of daily living. It comprises of 10 questions about daily living while the score is converted to percentage where 0% indicates no limitation in function while 50-100% indicates complete activity limitation. It has moderate test re-test reliability where ICC varies between 0.50 and 0.98, while it constructs a good validity.

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36) for quality of life | up to 12 weeks
  This survey quantifies the quality of life. It comprises of 36questions related to health, physical activity and psychology. It has shown to be reliable and a valid questionnaire.Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high quality of life.SF-36 scores range from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Misha Butt, MS*, Principal Investigator — Riphah International University
Locations (1):
- Noor Fatima Hospital, Dinga, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Genebra CVDS, Maciel NM, Bento TPF, Simeao SFAP, Vitta A. Prevalence and factors associated with neck pain: a population-based study. Braz J Phys Ther. 2017 Jul-Aug;21(4):274-280. doi: 10.1016/j.bjpt.2017.05.005. Epub 2017 May 20. PMID 28602744
- [Background] Childs JD, Cleland JA, Elliott JM, Teyhen DS, Wainner RS, Whitman JM, Sopky BJ, Godges JJ, Flynn TW; American Physical Therapy Association. Neck pain: Clinical practice guidelines linked to the International Classification of Functioning, Disability, and Health from the Orthopedic Section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2008 Sep;38(9):A1-A34. doi: 10.2519/jospt.2008.0303. Epub 2008 Sep 1. PMID 18758050
- [Background] Berg HE, Berggren G, Tesch PA. Dynamic neck strength training effect on pain and function. Arch Phys Med Rehabil. 1994 Jun;75(6):661-5. doi: 10.1016/0003-9993(94)90189-9. PMID 8002765
- [Background] Hrysomallis C. Neck Muscular Strength, Training, Performance and Sport Injury Risk: A Review. Sports Med. 2016 Aug;46(8):1111-24. doi: 10.1007/s40279-016-0490-4. PMID 26861960
- [Background] Lin IH, Chang KH, Liou TH, Tsou CM, Huang YC. Progressive shoulder-neck exercise on cervical muscle functions in middle-aged and senior patients with chronic neck pain. Eur J Phys Rehabil Med. 2018 Feb;54(1):13-21. doi: 10.23736/S1973-9087.17.04658-5. Epub 2017 Jul 17. PMID 28714658
- [Background] Conley MS, Stone MH, Nimmons M, Dudley GA. Specificity of resistance training responses in neck muscle size and strength. Eur J Appl Physiol Occup Physiol. 1997;75(5):443-8. doi: 10.1007/s004210050186. PMID 9189733
- [Background] Salo PK, Hakkinen AH, Kautiainen H, Ylinen JJ. Effect of neck strength training on health-related quality of life in females with chronic neck pain: a randomized controlled 1-year follow-up study. Health Qual Life Outcomes. 2010 May 14;8:48. doi: 10.1186/1477-7525-8-48. PMID 20465854
- [Background] Hakkinen A, Kautiainen H, Hannonen P, Ylinen J. Strength training and stretching versus stretching only in the treatment of patients with chronic neck pain: a randomized one-year follow-up study. Clin Rehabil. 2008 Jul;22(7):592-600. doi: 10.1177/0269215507087486. PMID 18586810
- [Background] Gallego-Sendarrubias GM, Rodriguez-Sanz D, Calvo-Lobo C, Martin JL. Efficacy of dry needling as an adjunct to manual therapy for patients with chronic mechanical neck pain: a randomised clinical trial. Acupunct Med. 2020 Aug;38(4):244-254. doi: 10.1136/acupmed-2018-011682. Epub 2020 Mar 23. PMID 32202124
- [Derived] Amjad M, Ur Rehman SS, Fatima G, Ikram M, Ghafoor S. Comparative effects of isometric and isotonic global neck muscles strengthening exercise programme on pain, range of motion, strength, function and quality of life in patients with chronic mechanical neck pain. J Pak Med Assoc. 2024 Oct;74(10):1843-1846. doi: 10.47391/JPMA.11378. PMID 39407381